CLINICAL TRIAL: NCT07266766
Title: An Open Label, Balanced, Randomized, Single Dose, Two Treatment, Two Sequence, Two Period, Two Way Crossover, Oral Bioequivalence Study of Test Product of Empagliflozin / Metformin 25 mg/ 1000 mg Extended-Release Tablet and Reference Product of Synjardy XR Tablets 25mg/1000mg in Healthy, Adult, Human Subjects Under Fed Condition.
Brief Title: Bioequivalence Study to Compare Empagliflozin / Metformin 25 mg/ 1000 mg Extended-Release Tablet Versus Synjardy XR Tablets 25mg/1000mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 25-VIN-0321
Record Dates: First submitted 2025-11-28; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin / Metformin HCl XR Tablets (Experimental): Empagliflozin / Metformin HCl XR 25 mg/ 1000 mg Tablets
  Interventions: Drug: Empagliflozin / Metformin HCl XR Tablets; Drug: Synjardy® XR (empagliflozin and metformin hydrochloride extended-release Tablets)
- Synjardy® XR (empagliflozin and metformin hydrochloride extended-release Tablets) (Active Comparator): Synjardy® XR (empagliflozin and metformin hydrochloride extended-release Tablets) 25 mg/1000 mg
  Interventions: Drug: Empagliflozin / Metformin HCl XR Tablets; Drug: Synjardy® XR (empagliflozin and metformin hydrochloride extended-release Tablets)

INTERVENTIONS:
Drug: Empagliflozin / Metformin HCl XR Tablets — One Empagliflozin / Metformin HCl XR 25 mg/ 1000 mg Tablets
Drug: Synjardy® XR (empagliflozin and metformin hydrochloride extended-release Tablets) — One Synjardy® XR (empagliflozin and metformin hydrochloride extended-release Tablets) 25 mg/1000 mg

SUMMARY:
An Open Label, Balanced, Randomized, Single dose, Two treatment, Two sequence, Two period, two way crossover, Oral Bioequivalence Study of test product of Empagliflozin / Metformin 25 mg/ 1000 mg Extended-Release Tablet and Reference product of Synjardy XR tablets 25mg/1000mg in Healthy, adult, human Subjects Under fed Condition.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 to 45 years (both inclusive).
* Subjects' weight within normal range according to normal values for Body Mass Index (between 18.5 to 30.0 kg/m2) (both inclusive) with minimum of 45 kg weight.
* Subjects with normal health as determined by personal medical history, clinical examination and laboratory examinations within Predefined site Normal range.
* Subjects having clinically acceptable 12-lead electrocardiogram (ECG).
* Subjects having clinically acceptable chest X-Ray (PA view), if taken.
* Subjects having negative urine screen for drugs of abuse (including amphetamines, barbiturates, benzodiazepines, marijuana, cocaine, and morphine).
* Subjects having negative urine alcohol test / breath alcohol test.
* Non-smoker.
* Subjects willing to adhere to the protocol requirements and to provide written informed consent.
* Subject with Creatinine Clearance ˃60 ml/min.
* For male Subjects:

Subjects willing to follow approved birth control methods (a double barrier method) for the duration of the study as judged by the investigator(s), such as (a double barrier method) condom with spermicide, Condom with diaphragm, or abstinence. Subjects willing to refrain from donating sperm during the study period - For Female Subjects: Female of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as intrauterine device (IUD), abstinence, bilateral tubal ligation or double barrier contraception, i.e., condom + diaphragm, condom + spermicidal or foam Postmenopausal for at least 1 year, or if less than 1 year, then following acceptable contraceptive measures as mentioned above

- Subjects having negative urine pregnancy test at screening and negative serum b-hCG pregnancy test on admission day of period 01 (only for female subjects).

Exclusion Criteria:

* Hypersensitivity to Empagliflozin and Metformin or related class of drugs or any of its excipients or heparin.
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological, urogenital or psychiatric disease or disorder.
* Any treatment which could bring about induction or inhibition of hepatic microsomal enzyme system within 30 days prior to admission in period 01.
* Presence of alcoholism or drug abuse.
* History or presence of asthma, urticaria or other significant allergic reactions.
* History or presence of significant gastric and/or duodenal ulceration.
* History or presence of significant thyroid disease, adrenal dysfunction, organic intracranial lesion such as pituitary tumor.
* History or presence of cancer or basal or squamous cell carcinoma.
* Difficulty with donating blood.
* Difficulty in swallowing solids dosage form like tablets or capsules.
* Use of any prescribed medication or OTC medication including vaccines, vitamins and herbal remedies during last 30 days prior to admission in period 01.
* Major illness within past 3 months.
* Volunteer who have donated blood (1 unit) or participation in a drug research study within past 90 days prior to the first dose of the study drug.
* Consumption of xanthine-containing products, tobacco containing products or alcohol or any alcohol containing products within 48.00 hours prior to admission in period 01.
* Consumption of grapefruit or grapefruit juice containing products within 72.00 hours prior to admission of period 01.
* Positive screening test for any one or more: HIV, Hepatitis B and Hepatitis C.
* History or presence of significant easy bruising or bleeding.
* History or presence of significant recent trauma.
* Subjects who have been on an abnormal diet (for whatever reason) during the four weeks preceding the study.
* History of any type of acute metabolic acidosis (such as lactic acidosis, diabetic ketoacidosis).
* History of Diabetic pre-coma.
* History of acute conditions with the potential to alter renal function such as: dehydration, severe infection, shock.
* History of disease which may cause tissue hypoxia (especially acute disease, or worsening of chronic disease) such as: decompensated heart failure, respiratory failure, recent myocardial infarction, shock.
* History of Hepatic impairment or acute alcohol intoxication.
* Female subjects who are currently breast feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-08-05 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
For Empagliflozin & Metformin; Maximum concentration obtained (Cmax) | 72 hours
  two-sides 90% CI for the test to reference ratio of the population means is within 80.00-125.00% for each of the Ln-transformed data Cmax
For Empagliflozin & Metformin; AUC from time 0 to last collection time (AUC0 - t) | 72 hours
  two-sides 90% CI for the test to reference ratio of the population means is within 80.00-125.00% for each of the Ln-transformed data AUC

SECONDARY OUTCOMES:
For Empagliflozin & Metformin; Time to reach maximum concentration Cmax (Tmax) | 72 hours
  Descriptive Statistics
For Empagliflozin & Metformin; AUC0-24 | 72 hours
  Descriptive Statistics

CONTACTS AND LOCATIONS:
Locations (1):
- Veeda Clinical Research Limited, Ahmedabad, Gujarat, India